CLINICAL TRIAL: NCT06353906
Title: A Phase 2 Clinical Study to Assess Efficacy of Induction Carboplatin/Paclitaxel + Pembrolizumab for Locoregionally Advanced Penile Cancer: PRIAM
Brief Title: Carboplatin/Paclitaxel + Pembrolizumab for Locoregionally Advanced Penile Cancer
Acronym: PRIAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N22APC
Record Dates: First submitted 2024-03-15; First posted 2024-04-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Urologic Neoplasms; Urogenital Neoplasms; Male Urogenital Diseases; Penile Cancer; Penile Squamous Cell Carcinoma; Locally Advanced Penile Carcinoma
MeSH Terms: conditions — Urologic Neoplasms; Urogenital Neoplasms; Male Urogenital Diseases; Penile Neoplasms | interventions — CP protocol; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction chemo-immunotherapy combination followed by consolidative surgical resection (Experimental): Patients receive three cycles of induction carboplatin+paclitaxel on days 1, 22 and 43, with two concurrent cycles of fixed-dose pembrolizumab on days 1 and 43.
  Within 3-9 weeks after the last cycle of induction chemo-immunotherapy, patients undergo complete resection of remaining tumor tissue.
  Patients start subsequent adjuvant immunotherapy with fixed-dose pembrolizumab for up to seven 6-week cycles between 3-9 weeks after surgery.
  Interventions: Drug: Carboplatin/Paclitaxel; Drug: Pembrolizumab; Procedure: Partial or total penectomy with inguinal and/or pelvic lymph node dissection

INTERVENTIONS:
Drug: Carboplatin/Paclitaxel — Induction: three cycles of intravenous carboplatin AUC5 (max 750 mg) and paclitaxel 175 mg/m2, during cycle 1, 2 and 3 (day 1, 22, 43)
  Other Names: CarboTaxol; PC
Drug: Pembrolizumab — Induction: two cycles of intravenous pembrolizumab 400 mg during cycle 1 and 3 (day 1 and 43)
  Adjuvant: up to seven cycles of fixed-dose intravenous pembrolizumab 400 mg, on day 1 every 6 weeks within 3-9 weeks after surgery
  Other Names: Keytruda
Procedure: Partial or total penectomy with inguinal and/or pelvic lymph node dissection — Resection of part or all of the penis with complete removal of suspect lymphnodes in the inguinal and/or pelvic area
  Other Names: Inguinal lymphadenectomy; groin dissection; PLND

SUMMARY:
This is a single-armed, single-centre, non-blinded phase II trial to assess efficacy of induction chemo-immunotherapy for resectable node-positive squamous cell carcinoma of the penis

DETAILED DESCRIPTION:
This is a phase II study in which fifty adult patients with cTxN1-3 locoregionally advanced squamous cell penile cancer (LRAPC), suitable for resection will be included. Patients with recurrence in lymph nodes are suitable for inclusion if they have not received prior systemic treatment. Patients with cN1 are only included in case of central nodal necrosis and/or an irregular nodal border, or node >3cm on CT. A maximum of 2 supraregional or distant metastases is allowed if local treatment (i.e. irradiation or resection) is feasible.

Patients will be treated with three 21-day cycles of induction chemotherapy, carboplatin AUC5 (max 750 mg) and paclitaxel 175 mg/m2, with additional fixed-dose 400mg pembrolizumab on the first and third cycle.

Response to induction therapy will be evaluated by CT scan, ca. 2 weeks after the last cycle.

Subsequent consolidative treatment will consist of surgical resection of all visible and/or suspected disease.

In 3-9 weeks after surgery, patients will enter the adjuvant phase, consisting of 7 cycles of pembrolizumab 400 mg every 6 weeks. Focused physical examination, registration of adverse-events and monitoring of, amongst others, TSH, FT4, liver enzymes via blood tests, is performed at the start of every cycle. End of treatment visit will be set 30 days after receiving the last cycle of pembrolizumab.

Disease status will be monitored by CT-scan at 3, 6, 9, 12, 18 and 24 months from resection, after which imaging will follow standard follow-up protocols. QoL will be assessed at 3,6,12, 18 and 24 months using using the EORTC QLQ-C30 questionnaire. Following 24 months after resection subsequent follow-up visits for survival and anti-cancer therapy will be planned every 6 months, until death, withdrawal of consent or the end of the study, whichever occurs first.

The primary endpoint is efficacy, defined as pathological complete response (pCR).

Secondary endpoints are grade 3-4 toxicity (by CTCAE 5.0), PFS and OS at 2 years after surgery, correlation of clinical endpoints (pCR, PFS, OS) with high-risk HPV (hrHPV) and PD-L1 immunohistochemistry, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Histologically confirmed diagnosis of squamous cell carcinoma of the penis.
3. Patients have one of the following disease stages:

   * cTxN2-3 or
   * cTxN1 in case of central nodal necrosis and/or an irregular nodal border, or node >3cm, or
   * Inguinal or pelvic lymph node recurrence that is potentially resectable. Any of the disease stages above, in combination with oligometastatic disease with a maximum of 2 distant metastases is allowed, as long as these metastases can be treated by resection or radiotherapy. This should be established in the multidisciplinary tumor board before enrolment.
4. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
5. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 14 days prior to the first dose of study intervention.
7. Have adequate organ function defined as: absolute neutrophil count (ANC) ≥1.5 10e9 /L, platelets ≥100 10e9/L; hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L; creatinine ≤1.5 × ULN OR GFR>30 ml/min as per Cockcroft-Gault formula in patients with creatinine levels > 1.5x institutional ULN; total bilirubin 1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN; AST (SGOT) and ALT (SGPT) ≤2.5 × ULN; International normalized ratio (INR), prothrombin time (PT) OR activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants. Specimens must be collected within 14 days prior to the start of study intervention.

Exclusion Criteria:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
2. Has received prior systemic anti-cancer therapy including investigational agents, or an investigational device, within 4 weeks prior to registration.
3. Has received prior radiotherapy within 4 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids.
4. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Exceptions: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded. Patients with low-risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
7. Has known active or treated CNS metastases and/or carcinomatous meningitis.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid). Patients with vitiligo, psoriasis or other mild skin disease can still be included.
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Human Immunodeficiency Virus (HIV) infection.
13. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and/or Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Hepatitis B and C screening tests are not required unless a patient has a known history of HBV or HCV infection. Participants must have completed curative anti-viral therapy at least 6 months prior to randomization.
14. Has not adequately recovered from major surgery or has ongoing surgical complications.
15. Major pelvic surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for the disease under study.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is expecting to father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2028-01-14 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Immediately after surgery
  Pathological complete response defined as pT0N0 in all evaluable patients

SECONDARY OUTCOMES:
Drug toxicity | Drug-related serious adverse events will be noted from day of registration until 90 days after the last protocol treatment/administration.
  Safety in terms of chemotherapy and immunotherapy-related adverse events of grade 3 or higher according to version 5.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) criteria.
Progression-free survival (PFS) | Through study completion, at a minimum of 24 months
  PFS is defined as time from start of therapy until an event.
  Events include:
  * Histologically or cytologically established recurrence after surgery
  * Omission of surgery as a result of progressive disease.
  * Unequivocal radiological progression. In case of equivocal results, radiological evaluation may continue. When unequivocal progression is established, the event date will be the first tumor assessment where new lesions were noted.
  * Switch to another systemic therapy. Note: in case a radiologically responding patient refuses surgery and elects other locoregional therapy (e.g. (chemo)radiotherapy), this is not considered a progression event.
  PFS will be estimated using the Kaplan-Meier method. The median PFS and 95% confidence interval will be reported.
Overall survival (OS) | Through study completion, at a minimum of 24 months
  OS is defined as the time between the date of enrollment and the date of death. OS will be estimated using the Kaplan-Meier method. The median OS and 95% confidence interval will be reported.
Assessment of correlation between clinical endpoints and tumor characteristics | Tumor tissue will be collected at baseline and during resection procedure. Clinical endpoints of pCR, PFS and OS will be determined as mentioned above
  Tumor tissue gathered from patients at baseline via biopsy and, in case of non complete response, at surgery will be tested via a comprehensive analysis of the tumor microenvironment (TME) using state of the art multiparameter techniques to determine the TME composition and activation status in responders vs non-responders. Additional analyses on clinical endpoints (i.e. pCR, PFS and OS) will be carried out between patient groups defined by tumor characteristics.
Tumor tissue HPV status in relation to treatment response | 12 weeks after last patient first visit
  HPV, or human papilloma virus, status of pre-treatment (baseline) tumor tissue will be determined. Tumor tissue will be tested for HPV status (present or not) to determine a possible (prior) infection with a "high-risk" HPV serotype. High-risk meaning a serotype associated with a higher risk for developing neoplasms. High-risk HPV status will be related to pCR, PFS and OS as they are described above. Baseline tumor tissue will be requested from a referring hospital or gathered from each individual patient during screening.
Tumor tissue PD-L1 expression in relation to treatment response | 12 weeks after last patient first visit
  PD-L1 expression of pre-treatment (baseline) tumor tissue will be determined. PD-L1 tumor proportion score (TPS; 0%-100%) will be assessed via immunohistochemical staining of tumor tissue. PD-L1 TPS ≥50% will be related to pCR, PFS and OS as they are described above. Baseline tumor tissue will be requested from a referring hospital or gathered from each individual patient during screening.
Evaluation of changes in patient reported outcome regarding Quality of Life (QoL) | From screening until end of treatment visit (30 days after last adjuvant treatment)
  QoL will be measured by the European Organization for the Research and Treatement of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) in all patients who were registered for the study and started treatment. This questionnaire will be used to evaluate changes from baseline in QoL, with patient-reported QoL scored in various domains on a scale of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel S. van der Heijden, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- UZ Leuven, Leuven, Belgium
- NKI-AVL, Amsterdam, North Holland, Netherlands